CLINICAL TRIAL: NCT00286793
Title: An Open-label, Multicenter, Phase I/II Study of AT-101 in Combination With Docetaxel and Prednisone in Men With Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Safety and Efficacy Study of AT-101 in Combination With Docetaxel and Prednisone in Men With HRPC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Kimberli Brill, Associate Director, Clinical Development, Ascenta Therapeutics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-202
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
Keywords: at-101; at101; cancer; hormone refractory; prostate; docetaxel; prednisone
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIngle Arm Study of AT-101 in combination with Docetaxel (Experimental)
  Interventions: Drug: AT-101

INTERVENTIONS:
Drug: AT-101 — Oral

SUMMARY:
This is an open-label, multicenter Phase I/II study to evaluate the safety and efficacy of AT-101 in combination with docetaxel and prednisone in men with hormone-refractory prostate cancer that are either chemotherapy naive or have received and progressed on a docetaxel containing regimen,

ELIGIBILITY:
Inclusion Criteria:

1. Rising prostate specific antigen (PSA) despite castrate levels of testosterone due to orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist therapy.
2. Patients must have metastatic disease by bone scan, computed tomography (CT) scan, or magnetic resonance imaging (MRI).
3. ECOG performance status 0 or 1
4. Adequate hematologic function
5. Adequate liver and renal function
6. Able to swallow and retain oral medication.
7. Patients enrolled into Cohort B must have documented progression of disease during treatment with a docetaxel-containing regimen by meeting one or more of the following criteria- rising PSA, progression of disease per RECIST, or >2 new lesions on bone scan.
8. Patients enrolled into Cohort B must have received at least two cycles of docetaxel. Minimum doses of prior docetaxel permitted are 60 mg/m2 on a q 3 week schedule or 20 mg/m2 on a weekly schedule.
9. At least 4 weeks since prior flutamide, megestrol, ketoconazole, and radiotherapy, and at least 6 weeks since prior bicalutamide or nilutamide.

Exclusion Criteria:

1. Patients enrolled into Cohort A must not have received prior chemotherapy for HRPC.
2. Known history of or clinical evidence of central nervous system (CNS) metastases.
3. Active secondary malignancy or history of other malignancy within the last 5 years.
4. Prior history of radiation therapy to > 25% of the bone marrow
5. Peripheral neuropathy of > Grade 2
6. Uncontrolled concurrent illness
7. Failure to recover fully, as judged by the investigator, from prior surgical procedures.
8. Concurrent anti-cancer therapy other than docetaxel and prednisone.
9. Patients must not be receiving concurrent anti-androgen hormonal therapy for HRPC (LHRH therapies are acceptable to maintain castrate levels of testosterone)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety of AT-101 in combination with docetaxel and prednisone | 12 months

SECONDARY OUTCOMES:
Preliminary efficacy of AT-101 in combination with docetaxel and prednisone | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Ascenta Therapeutics, Inc.
Locations (13):
- United States (13):
  - Hot Springs, Arkansas
  - Fort Meyers, Florida
  - Chicago, Illinois
  - Fridley, Minnesota
  - Albuquerque, New Mexico
  - Syracuse, New York
  - Wilmington, North Carolina
  - Portland, Oregon
  - Hilton Head Island, South Carolina
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Richardson, Texas